CLINICAL TRIAL: NCT04256824
Title: Triclosan-antibacterial Sutures Efficacy on the Incidence of Surgical Site Infection in Clean-contaminated Wounds; Multi-center, Double Blind, Randomized Study
Brief Title: Triclosan-antibacterial Sutures Efficacy on the Incidence of Surgical Site Infection in Clean-contaminated Wounds
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ClinAmygate (Other)
Collaborators: Misr University for Science and Technology (Other); Al Safwa Hospital (Unknown); Al Zohour Hospital (Unknown); Al-Menia Univeristy Hospital (Unknown); MSKMC Univeristy Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR2019-27
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Surgical Site Infection; Surgical Wound; Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound | interventions — Triclosan; Polyglactin 910

STUDY DESIGN:
Intervention Model Description: randomized-controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Coated Polyglactin 910 with Triclosan (Experimental): Coated vicryl plus
  Interventions: Drug: coated vicryl plus
- Coated Polyglactin 910 without Triclosan (Active Comparator): Coated vicryl
  Interventions: Drug: Vicryl

INTERVENTIONS:
Drug: coated vicryl plus — Coated Polyglactin 910 with Triclosan (coated vicryl plus)
  Other Names: Coated Polyglactin 910 with Triclosan
  Arms: Coated Polyglactin 910 with Triclosan
Drug: Vicryl — Coated Polyglactin 910 without Triclosan (vicryl)
  Other Names: Coated Polyglactin 910 without Triclosan
  Arms: Coated Polyglactin 910 without Triclosan

SUMMARY:
Comparing the incidence of SSI in cases using coated Polyglactin 910 suture with Triclosan and cases using Polyglactin 910 suture without Triclosan in clean-contaminated wound surgery

DETAILED DESCRIPTION:
Comparing the incidence of surgical site infection (SSI) in cases using coated Polyglactin 910 suture with Triclosan and cases using Polyglactin 910 suture without Triclosan in clean-contaminated wound surgery. Also, comparing the post hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-75
* clean-contaminated wound surgery

Exclusion Criteria:

* Patient has immunodeficiency disorder.
* Patient receiving anti-cancer / immunosuppressive therapy.
* Patients with established pre-operative infection whether community acquired or hospital acquired either at / remote from the operative site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 30 days
  Incidence of surgical site infection within 30 days

SECONDARY OUTCOMES:
Hospital stay | 30 days
  duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, Diploma, Study Director — ClinAmygate
Locations (1):
- Misr Univeristy for Science and Technology Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmed I, Boulton AJ, Rizvi S, Carlos W, Dickenson E, Smith NA, Reed M. The use of triclosan-coated sutures to prevent surgical site infections: a systematic review and meta-analysis of the literature. BMJ Open. 2019 Sep 3;9(9):e029727. doi: 10.1136/bmjopen-2019-029727. PMID 31481559